CLINICAL TRIAL: NCT02685254
Title: Effects of Structured Skills Training Group in Treatment of ADHD in Adults: a Controlled Multicentre Study
Brief Title: Effects of Structured Skills Training Group in Treatment of ADHD in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Haukeland University Hospital (Other); Oslo University Hospital (Other); The Hospital of Vestfold (Other)
Responsible Party: Principal Investigator, Mats Fredriksen, Chief Attending Physician, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/1523 A
Record Dates: First submitted 2016-02-12; First posted 2016-02-18 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: Group Therapy; Structured Skills Training; Dialectic Behavioural Therapy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Initial group therapy (Experimental): 'Structural skills training group' - Start up with weekly structured skills training group for 14 weeks supplemented by homework training
  Interventions: Behavioral: Structural skills training group
- Initial control condition (Other): Treatment as usual/clinical management the first 15 weeks pending deferred start of group therapy (partially cross-over)
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Structural skills training group — Weekly 2-hours sessions for 14 weeks follow the Norwegian translation of the Swedish version of the ADHD skills training manual/workbook (Hesslinger 2010; Hirvikoski 2011; Morgensterns 2015) which is based on an adaption of Marsha Linehan's dialectical behavior therapy (DBT) for borderline personality disorder into a group-based skills training program for adults with ADHD (Hesslinger 2002; Philipsen 2007). The groups embrace 7 - 10 participants, and two group leaders trained in group therapy, cognitive-behavioral treatment or DBT. Each session contains an initial short repetition and feedback on the previous session, followed by review of the homework during the first hour. After a break, a new topic with exercises and homework for the following week is introduced.
  Other Names: Dialectic behavioural group therapy
  Arms: Initial group therapy
Other: Treatment as usual — Treatment as usual includes clinical management and/or medication, and or supportive counselling by physician or nurse
  Arms: Initial control condition

SUMMARY:
This study aims to examine if structured skills training group therapy for ADHD in adults has beneficial effects superior to 'treatment as usual' including medication in a controlled outpatient setting on clinically relevant outcomes including symptoms, functioning and quality of life measures.

The trial is designed as a multicenter randomized controlled, parallel group study. Patients are randomized into 1 of 2 treatment arms with 14-week duration: one arm with initial intervention by structured skills training groups by weekly sessions or one with control condition (treatment as usual). Then after 15 weeks patients in the control condition arm are switched to the active intervention by 14 weeks of structured group therapy. All patients are assessed for defined outcomes after six months.

DETAILED DESCRIPTION:
Background: The focus in recent years on evidence for non-pharmacological treatment in adults with ADHD raises the question of potential effects of structured group therapy. Structured skills training groups have shown beneficial effects in some studies in an outpatient psychiatric context by reduction in ADHD symptoms in individuals who remained stable regarding medication status.

Aims: The main objective for the trial is to investigate the potential effects of structured skills training groups in a clinically relevant but still controlled setting on broader outcomes including both symptomatic, functional and health related quality of life measures.

Methods/Design: The trial is designed as a multicenter randomized controlled parallel group design. At each outpatient site the enrolled patients are randomized into two groups for either Group 1 (G1) with start of weekly treatment in active structured skills training group lasting for 14 weeks or allocated to Group 2 (G2) with treatment as usual/clinical management and with 15 weeks delayed start of their group treatment for comparison wth patients in the other arm. Those patients in the control condition arm receiving treatment as usual or clinical management of individual patients (G2), are thereafter switched to active structured skills training group therapy.All patients are followed up after six months with assessments of primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADHD according to the Diagnostic and Statistical Manual of Mental Disorders, 4th. Edition (DSM-IV) persisting in adulthood

Exclusion Criteria:

* Any psychotic disorder
* Recently suicidal behaviour
* Substance or alcohol abuse or dependence within three months prior to screening for inclusion
* Pervasive developmental disorder
* Intellectual disability
* Seizures or any neurological diseases causing mental handicap

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Behaviour Rating Inventory of Executive Functions (BRIEF) | two years
  Change in executive function impairments

SECONDARY OUTCOMES:
Adult ADHD self-report scale (ASRSv1.1), 18 items version | two years
  Change in ADHD symptoms
Beck Depression Inventory (BDI) | two years
  Change in depressive symptoms
Beck Anxiety Inventory (BAI) | two years
  Change in anxiety symptoms
Weiss Functional Impairment Rating Scale, self-report (WIFRS) | two years
  Change in functional impairments
Global Assessment of functioning (GAF) | two years
  Change in global symptoms and functioning
Adult ADHD Quality of Life Scale (AAQoL) | two years
  Change in quality of life
Difficulties in Emotion Regulation Scale (DERS) | two years
  Change in emotional regulation
Safety issue - Monitoring of adverse events | two years
  Monitoring of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ellen K Munkhaugen, MSED, Study Director — Hospital of Oslo
Locations (1):
- Division of Mental Health and Addiction, Vestfold Hospital Trust, Tønsberg, Norway

IPD SHARING:
Plan to Share IPD: No
Data from each site will be anonymised in the final analyses

REFERENCES:
- [Background] Philipsen A, Richter H, Peters J, Alm B, Sobanski E, Colla M, Munzebrock M, Scheel C, Jacob C, Perlov E, Tebartz van Elst L, Hesslinger B. Structured group psychotherapy in adults with attention deficit hyperactivity disorder: results of an open multicentre study. J Nerv Ment Dis. 2007 Dec;195(12):1013-9. doi: 10.1097/NMD.0b013e31815c088b. PMID 18091195
- [Background] Philipsen A, Graf E, Jans T, Matthies S, Borel P, Colla M, Gentschow L, Langner D, Jacob C, Gross-Lesch S, Sobanski E, Alm B, Schumacher-Stien M, Roesler M, Retz W, Retz-Junginger P, Kis B, Abdel-Hamid M, Heinrich V, Huss M, Kornmann C, Burger A, van Elst LT, Berger M. A randomized controlled multicenter trial on the multimodal treatment of adult attention-deficit hyperactivity disorder: enrollment and characteristics of the study sample. Atten Defic Hyperact Disord. 2014 Mar;6(1):35-47. doi: 10.1007/s12402-013-0120-z. Epub 2013 Oct 17. PMID 24132867
- [Background] Philipsen A, Jans T, Graf E, Matthies S, Borel P, Colla M, Gentschow L, Langner D, Jacob C, Gross-Lesch S, Sobanski E, Alm B, Schumacher-Stien M, Roesler M, Retz W, Retz-Junginger P, Kis B, Abdel-Hamid M, Heinrich V, Huss M, Kornmann C, Burger A, Perlov E, Ihorst G, Schlander M, Berger M, Tebartz van Elst L; Comparison of Methylphenidate and Psychotherapy in Adult ADHD Study (COMPAS) Consortium. Effects of Group Psychotherapy, Individual Counseling, Methylphenidate, and Placebo in the Treatment of Adult Attention-Deficit/Hyperactivity Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2015 Dec;72(12):1199-210. doi: 10.1001/jamapsychiatry.2015.2146. PMID 26536057
- [Background] Hirvikoski T, Waaler E, Alfredsson J, Pihlgren C, Holmstrom A, Johnson A, Ruck J, Wiwe C, Bothen P, Nordstrom AL. Reduced ADHD symptoms in adults with ADHD after structured skills training group: results from a randomized controlled trial. Behav Res Ther. 2011 Mar;49(3):175-85. doi: 10.1016/j.brat.2011.01.001. Epub 2011 Jan 14. PMID 21295767
- [Background] Morgensterns E, Alfredsson J, Hirvikoski T. Structured skills training for adults with ADHD in an outpatient psychiatric context: an open feasibility trial. Atten Defic Hyperact Disord. 2016 Jun;8(2):101-11. doi: 10.1007/s12402-015-0182-1. Epub 2015 Sep 26. PMID 26410823
- [Background] Hesslinger B, Tebartz van Elst L, Nyberg E, Dykierek P, Richter H, Berner M, Ebert D. Psychotherapy of attention deficit hyperactivity disorder in adults--a pilot study using a structured skills training program. Eur Arch Psychiatry Clin Neurosci. 2002 Aug;252(4):177-84. doi: 10.1007/s00406-002-0379-0. PMID 12242579
- [Derived] Halmoy A, Ring AE, Gjestad R, Moller M, Ubostad B, Lien T, Munkhaugen EK, Fredriksen M. Dialectical behavioral therapy-based group treatment versus treatment as usual for adults with attention-deficit hyperactivity disorder: a multicenter randomized controlled trial. BMC Psychiatry. 2022 Nov 28;22(1):738. doi: 10.1186/s12888-022-04356-6. PMID 36443712